CLINICAL TRIAL: NCT00867841
Title: A Polymerase Chain Reaction-based Method to Improve Antibiotic Prescribing for Children and Adolescents With Community-Acquired Pneumonia - a Pilot Study
Brief Title: A Polymerase Chain Reaction (PCR) - Based Method to Improve Antibiotic Prescribing for Pneumonia
Status: Withdrawn | Type: Observational
Why Stopped: funding issues and procedural problems
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: CHEO-ID-001
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Pneumonia
Keywords: pneumonia, community-acquired; polymerase chain reaction; pneumococcus; mycoplasma; chlamydophila; anti-bacterial agents
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia; Mycoplasma Infections; Chlamydia Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasopharyngeal swabs blood samples (for pneumococcal PCR)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pneumonia: Children diagnosed with community-acquired pneumonia by the emergency department physician
  Interventions: Procedure: nasopharyngeal swab

INTERVENTIONS:
Procedure: nasopharyngeal swab — PCR of NP swab for Mycoplasma, Chlamydophila, pneumococcus, pneumococcus macrolide resistance genes.

SUMMARY:
Pneumonia, or lung infection, is usually treated with antibiotics targeted against the organisms that the physician guesses are causing the problem. The determination of the exact cause of a patient's pneumonia is difficult. The problem is that the two major causes of community-acquired pneumonia are not easily distinguished on clinical grounds and are best treated by different antibiotics. The investigators hypothesize that antibiotic therapy can be targeted and improved by doing polymerase chain reaction (PCR) testing of nose swabs to identify probable implicated organisms and their antibiotic resistance patterns. This pilot study will be important to ensure that the laboratory testing is functional and that the emergency department-laboratory communication is optimal prior to doing a full-fledged randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* presumed community-acquired pneumonia as diagnosed by the attending emergency department physician

Exclusion Criteria:

* age > 6 months
* immunodeficiency (primary, advanced HIV)
* cystic fibrosis
* malignancy
* known cardiac or lung defects
* bronchiectasis
* previous pneumonia or lung abscess in past 6 months
* conditions requiring treatment with immune suppressants

Min Age: 180 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: children with community-acquired pneumonia presenting to the Children's Hospital of Eastern Ontario emergency department
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Pernica, MD, Principal Investigator — Children's Hospital of Eastern Ontario/University of Ottawa; Robert Slinger, MD, Study Director — Children's Hospital of Eastern Ontario/University of Ottawa
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Esposito S, Bosis S, Cavagna R, Faelli N, Begliatti E, Marchisio P, Blasi F, Bianchi C, Principi N. Characteristics of Streptococcus pneumoniae and atypical bacterial infections in children 2-5 years of age with community-acquired pneumonia. Clin Infect Dis. 2002 Dec 1;35(11):1345-52. doi: 10.1086/344191. Epub 2002 Nov 13. PMID 12439797
- [Background] Michelow IC, Olsen K, Lozano J, Rollins NK, Duffy LB, Ziegler T, Kauppila J, Leinonen M, McCracken GH Jr. Epidemiology and clinical characteristics of community-acquired pneumonia in hospitalized children. Pediatrics. 2004 Apr;113(4):701-7. doi: 10.1542/peds.113.4.701. PMID 15060215
- [Background] Tsolia MN, Psarras S, Bossios A, Audi H, Paldanius M, Gourgiotis D, Kallergi K, Kafetzis DA, Constantopoulos A, Papadopoulos NG. Etiology of community-acquired pneumonia in hospitalized school-age children: evidence for high prevalence of viral infections. Clin Infect Dis. 2004 Sep 1;39(5):681-6. doi: 10.1086/422996. Epub 2004 Aug 13. PMID 15356783
- [Background] Juven T, Mertsola J, Waris M, Leinonen M, Meurman O, Roivainen M, Eskola J, Saikku P, Ruuskanen O. Etiology of community-acquired pneumonia in 254 hospitalized children. Pediatr Infect Dis J. 2000 Apr;19(4):293-8. doi: 10.1097/00006454-200004000-00006. PMID 10783017
- [Background] Munoz-Almagro C, Jordan I, Gene A, Latorre C, Garcia-Garcia JJ, Pallares R. Emergence of invasive pneumococcal disease caused by nonvaccine serotypes in the era of 7-valent conjugate vaccine. Clin Infect Dis. 2008 Jan 15;46(2):174-82. doi: 10.1086/524660. PMID 18171247
- [Background] Hicks LA, Harrison LH, Flannery B, Hadler JL, Schaffner W, Craig AS, Jackson D, Thomas A, Beall B, Lynfield R, Reingold A, Farley MM, Whitney CG. Incidence of pneumococcal disease due to non-pneumococcal conjugate vaccine (PCV7) serotypes in the United States during the era of widespread PCV7 vaccination, 1998-2004. J Infect Dis. 2007 Nov 1;196(9):1346-54. doi: 10.1086/521626. Epub 2007 Oct 4. PMID 17922399
- [Background] Korppi M, Heiskanen-Kosma T, Kleemola M. Incidence of community-acquired pneumonia in children caused by Mycoplasma pneumoniae: serological results of a prospective, population-based study in primary health care. Respirology. 2004 Mar;9(1):109-14. doi: 10.1111/j.1440-1843.2003.00522.x. PMID 14982611
- [Background] Chiang WC, Teoh OH, Chong CY, Goh A, Tang JP, Chay OM. Epidemiology, clinical characteristics and antimicrobial resistance patterns of community-acquired pneumonia in 1702 hospitalized children in Singapore. Respirology. 2007 Mar;12(2):254-61. doi: 10.1111/j.1440-1843.2006.01036.x. PMID 17298459
- [Background] Byington CL, Spencer LY, Johnson TA, Pavia AT, Allen D, Mason EO, Kaplan S, Carroll KC, Daly JA, Christenson JC, Samore MH. An epidemiological investigation of a sustained high rate of pediatric parapneumonic empyema: risk factors and microbiological associations. Clin Infect Dis. 2002 Feb 15;34(4):434-40. doi: 10.1086/338460. Epub 2002 Jan 3. PMID 11797168
- [Background] Eastham KM, Freeman R, Kearns AM, Eltringham G, Clark J, Leeming J, Spencer DA. Clinical features, aetiology and outcome of empyema in children in the north east of England. Thorax. 2004 Jun;59(6):522-5. doi: 10.1136/thx.2003.016105. PMID 15170039
- [Background] Thomson AH, Hull J, Kumar MR, Wallis C, Balfour Lynn IM. Randomised trial of intrapleural urokinase in the treatment of childhood empyema. Thorax. 2002 Apr;57(4):343-7. doi: 10.1136/thorax.57.4.343. PMID 11923554
- [Background] Shah SS, Alpern ER, Zwerling L, McGowan KL, Bell LM. Risk of bacteremia in young children with pneumonia treated as outpatients. Arch Pediatr Adolesc Med. 2003 Apr;157(4):389-92. doi: 10.1001/archpedi.157.4.389. PMID 12695236
- [Background] Johansson N, Kalin M, Giske CG, Hedlund J. Quantitative detection of Streptococcus pneumoniae from sputum samples with real-time quantitative polymerase chain reaction for etiologic diagnosis of community-acquired pneumonia. Diagn Microbiol Infect Dis. 2008 Mar;60(3):255-61. doi: 10.1016/j.diagmicrobio.2007.10.011. Epub 2007 Nov 26. PMID 18036762
- [Background] Lahti E, Mertsola J, Kontiokari T, Eerola E, Ruuskanen O, Jalava J. Pneumolysin polymerase chain reaction for diagnosis of pneumococcal pneumonia and empyema in children. Eur J Clin Microbiol Infect Dis. 2006 Dec;25(12):783-9. doi: 10.1007/s10096-006-0225-9. PMID 17089094
- [Background] Le Monnier A, Carbonnelle E, Zahar JR, Le Bourgeois M, Abachin E, Quesne G, Varon E, Descamps P, De Blic J, Scheinmann P, Berche P, Ferroni A. Microbiological diagnosis of empyema in children: comparative evaluations by culture, polymerase chain reaction, and pneumococcal antigen detection in pleural fluids. Clin Infect Dis. 2006 Apr 15;42(8):1135-40. doi: 10.1086/502680. Epub 2006 Mar 7. PMID 16575731
- [Background] Stralin K, Backman A, Holmberg H, Fredlund H, Olcen P. Design of a multiplex PCR for Streptococcus pneumoniae, Haemophilus influenzae, Mycoplasma pneumoniae and Chlamydophila pneumoniae to be used on sputum samples. APMIS. 2005 Feb;113(2):99-111. doi: 10.1111/j.1600-0463.2005.apm1130203.x. PMID 15723684
- [Background] Stralin K, Tornqvist E, Kaltoft MS, Olcen P, Holmberg H. Etiologic diagnosis of adult bacterial pneumonia by culture and PCR applied to respiratory tract samples. J Clin Microbiol. 2006 Feb;44(2):643-5. doi: 10.1128/JCM.44.2.643-645.2006. PMID 16455935
- [Background] Dagan R, Shriker O, Hazan I, Leibovitz E, Greenberg D, Schlaeffer F, Levy R. Prospective study to determine clinical relevance of detection of pneumococcal DNA in sera of children by PCR. J Clin Microbiol. 1998 Mar;36(3):669-73. doi: 10.1128/JCM.36.3.669-673.1998. PMID 9508293
- [Background] Kee C, Palladino S, Kay I, Pryce TM, Murray R, Rello J, Gallego M, Lujan M, Munoz-Almagro C, Waterer GW. Feasibility of real-time polymerase chain reaction in whole blood to identify Streptococcus pneumoniae in patients with community-acquired pneumonia. Diagn Microbiol Infect Dis. 2008 May;61(1):72-5. doi: 10.1016/j.diagmicrobio.2007.12.011. Epub 2008 Jan 24. PMID 18221851
- [Background] Rouphael NG, Atwell-Melnick N, Longo D, Whaley M, Carlone GM, Sampson JS, Ades EW. A real-time polymerase chain reaction for the detection of Streptococcus pneumoniae in blood using a mouse model: a potential new "gold standard". Diagn Microbiol Infect Dis. 2008 Sep;62(1):23-5. doi: 10.1016/j.diagmicrobio.2008.06.002. Epub 2008 Jul 14. PMID 18621498
- [Background] Harris KA, Turner P, Green EA, Hartley JC. Duplex real-time PCR assay for detection of Streptococcus pneumoniae in clinical samples and determination of penicillin susceptibility. J Clin Microbiol. 2008 Aug;46(8):2751-8. doi: 10.1128/JCM.02462-07. Epub 2008 Jun 18. PMID 18562586
- [Background] Ho PL, Wong RC, Chow FK, Cheung MY, Wong SS, Yam WC, Que TL. Application of a multiplex pbp2b and pbp2x PCR for prediction of penicillin resistance in Streptococcus pneumoniae. J Antimicrob Chemother. 2004 May;53(5):890-1. doi: 10.1093/jac/dkh216. Epub 2004 Apr 8. No abstract available. PMID 15073164
- [Background] Fukushima KY, Yanagihara K, Hirakata Y, Sugahara K, Morinaga Y, Kohno S, Kamihira S. Rapid identification of penicillin and macrolide resistance genes and simultaneous quantification of Streptococcus pneumoniae in purulent sputum samples by use of a novel real-time multiplex PCR assay. J Clin Microbiol. 2008 Jul;46(7):2384-8. doi: 10.1128/JCM.00051-08. Epub 2008 May 7. PMID 18463207
- [Background] Saukkoriipi A, Kaijalainen T, Kuisma L, Ojala A, Leinonen M. Isolation of pneumococcal DNA from nasopharyngeal samples for real-time, quantitative PCR: comparison of three methods. Mol Diagn. 2003;7(1):9-15. doi: 10.1007/BF03260015. PMID 14529315
- [Background] Normann E, Gnarpe J, Gnarpe H, Wettergren B. Chlamydia pneumoniae in children attending day-care centers in Gavle, Sweden. Pediatr Infect Dis J. 1998 Jun;17(6):474-8. doi: 10.1097/00006454-199806000-00007. PMID 9655537
- [Background] O'Brien KL, Nohynek H; World Health Organization Pneumococcal Vaccine Trials Carriage Working Group. Report from a WHO Working Group: standard method for detecting upper respiratory carriage of Streptococcus pneumoniae. Pediatr Infect Dis J. 2003 Feb;22(2):e1-11. doi: 10.1097/01.inf.0000049347.42983.77. PMID 12586987